CLINICAL TRIAL: NCT02600897
Title: A Phase Ib/II Study Evaluating the Safety and Efficacy of Obinutuzumab in Combination With Polatuzumab Vedotin and Lenalidomide in Patients With Relapsed or Refractory Follicular Lymphoma and Rituximab in Combination With Polatuzumab Vedotin and Lenalidomide in Patients With Relapsed or Refractory Diffuse Large B-Cell Lymphoma
Brief Title: A Study of Obinutuzumab, Polatuzumab Vedotin, and Lenalidomide in Relapsed or Refractory Follicular Lymphoma (FL) and Rituximab in Combination With Polatuzumab Vedotin and Lenalidomide in Relapsed or Refractory Diffuse Large B-Cell Lymphoma (DLBCL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: GO29834; 2015-001999-22 (EudraCT Number)
Record Dates: First submitted 2015-11-03; First posted 2015-11-09 (Estimated); Results first posted 2023-12-26 (Actual); Last update posted 2023-12-26 (Actual); Status verified 2023-12

CONDITIONS: Relapsed or Refractory Follicular Lymphoma, Relapsed or Refractory Diffuse Large B-Cell Lymphoma
MeSH Terms: conditions — Recurrence; Lymphoma, Follicular; Lymphoma, Large B-Cell, Diffuse | interventions — Lenalidomide; obinutuzumab; polatuzumab vedotin; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Dose-escalation Cohort: FL (Experimental): Participants with R/R FL will receive 6 months of induction treatment with polatuzumab vedotin and lenalidomide at escalating doses to identify the recommended Phase 2 dose (RP2D) for polatuzumab vedotin and lenalidomide when combined with a fixed dose of obinutuzumab. Those who achieve CR, PR, or SD at the EOI (6-8 weeks after Day 1 of Cycle 6) will be eligible to receive a 24-month maintenance regimen consisting of lenalidomide and obinutuzumab, to be initiated 8 weeks after Day 1 of Cycle 6 (induction cycle).
  Interventions: Drug: Lenalidomide; Drug: Obinutuzumab; Drug: Polatuzumab Vedotin
- Dose-escalation Cohort: DLBCL (Experimental): Participants with R/R DLBCL will receive 6 months of induction treatment with fixed dose of polatuzumab vedotin and rituximab along with dose escalating lenalidomide. Lenalidomide will be administered at escalating doses to identify the recommended Phase 2 dose (RP2D) for lenalidomide. Those who achieve CR and PR at the EOI (6-8 weeks after Day 1 of Cycle 6) will be eligible to receive a 6-month consolidation regimen consisting of lenalidomide and rituximab, to be initiated 8 weeks after Day 1 of Cycle 6 (induction cycle).
  Interventions: Drug: Lenalidomide; Drug: Polatuzumab Vedotin; Drug: Rituximab
- Expansion Cohort: FL (Experimental): Participants with R/R FL who received induction treatment with polatuzumab vedotin and lenalidomide, in addition to obinutuzumab and achieved CR, PR, or SD at the EOI (6-8 weeks after Day 1 of Cycle 6) will receive a 24-months maintenance regimen consisting of lenalidomide and obinutuzumab for first 12 months followed by obinutuzumab treatment for next 12 months. Post-induction therapy will start 8 weeks after Cycle 6 Day 1.
  Interventions: Drug: Lenalidomide; Drug: Obinutuzumab
- Expansion Cohort: DLBCL (Experimental): Participants with R/R DLBCL who received induction treatment with polatuzumab vedotin and lenalidomide in addition to rituximab and achieved CR or PR at the EOI (6-8 weeks after Day 1 of Cycle 6) will receive a 6-month consolidation regimen consisting of lenalidomide and rituximab. Post-induction therapy will start 8 weeks after Cycle 6 Day 1.
  Interventions: Drug: Lenalidomide; Drug: Rituximab

INTERVENTIONS:
Drug: Lenalidomide — All participants will receive lenalidomide oral capsules at doses of 10, 15, or 20 milligrams (mg) on Days 1 to 21 of each 28-day cycle for up to 6 Cycles in dose escalation phase followed by post-induction treatment at a dose of 10 mg once daily on Days 1 to 21 of each subsequent 28-day cycle. Post-induction lenalidomide may continue for up to 12 months until disease progression or unacceptable toxicity for participants with R/R FL and up to 6 months until disease progression or unacceptable toxicity for participants with R/R DLBCL.
Drug: Obinutuzumab — Participants will receive a fixed dose of obinutuzumab, 1000 mg via intravenous (IV) infusion to be given on Days 1, 8 and 15 of Cycle 1 and on Day 1 of Cycles 2 to 6 followed by post-induction treatment at a dose of 1000 mg via IV infusion on Day 1 of every other month for up to 24 months until disease progression or unacceptable toxicity.
  Arms: Dose-escalation Cohort: FL; Expansion Cohort: FL
Drug: Polatuzumab Vedotin — Participants with R/R FL will receive polatuzumab vedotin via IV infusion at doses of 1.4 or 1.8 milligrams per kilogram (mg/kg) on Day 1 of each 28-day cycle for up to 6 months during induction treatment. Participants wit R/R DLBCL will receive polatuzumab vedotin via IV infusion at dose 1.8 mg/kg on Day 1 of each 28-day cycle for up to 6 months during induction treatment.
  Arms: Dose-escalation Cohort: DLBCL; Dose-escalation Cohort: FL
Drug: Rituximab — Participants will receive a fixed dose of rituximab, 375 mg/m^2 via intravenous (IV) infusion to be given on Days 1 of Cycle 1 to 6 followed by post-induction treatment at a dose of 375 mg/m^2 via IV infusion on Day 1 of every other month for up to 6 months, until disease progression or unacceptable toxicity.
  Arms: Dose-escalation Cohort: DLBCL; Expansion Cohort: DLBCL

SUMMARY:
This study will evaluate the safety, efficacy, and pharmacokinetics of induction treatment with obinutuzumab, polatuzumab vedotin, and lenalidomide in participants with relapsed or refractory (R/R) follicular lymphoma (FL) and rituximab in combination with polatuzumab vedotin and lenalidomide in participants with R/R diffuse large B-cell lymphoma (DLBCL), followed by post-induction treatment with obinutuzumab in combination with lenalidomide in participants with FL who achieve a complete response (CR), partial response (PR), or stable disease (SD) at end of induction (EOI) and post-induction treatment with rituximab plus lenalidomide in participants with DLBCL who achieve a CR or PR at EOI.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to (>/=) 18 years
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* For obinutuzumab in combination with polatuzumab vedotin and lenalidomide (G + Pola + Len) treatment group: R/R FL after treatment with at least one prior chemoimmunotherapy regimen that included an anti-CD20 monoclonal antibody and for which no other more appropriate treatment option exists as determined by the investigator
* For rituximab in combination with polatuzumab vedotin and lenalidomide (R + Pola + Len) treatment group: R/R DLBCL after treatment with at least one prior chemoimmunotherapy regimen that included an anti-CD20 monoclonal antibody in patients who are not eligible for autologous stem-cell transplantation or who have experienced disease progression following treatment with high-dose chemotherapy plus autologous stem-cell transplantation
* Histologically documented CD20-positive B-cell lymphoma as determined by the local laboratory
* fluorodeoxyglucose (FDG)-avid lymphoma (i.e., positron emission tomography (PET)-positive lymphoma)
* At least one bi-dimensionally measurable lesion
* Agreement to remain abstinent or use adequate contraception, among women or men of childbearing potential

Exclusion Criteria:

* Grade 3b follicular lymphoma
* History of transformation of indolent disease to diffuse large B-cell lymphoma (DLBCL)
* Known CD20-negative status at relapse or progression
* Central nervous system (CNS) lymphoma or leptomeningeal infiltration
* Prior allogeneic stem-cell transplantation (SCT), or autologous SCT within 100 days prior to Day 1 of Cycle 1
* Current use of systemic immunosuppressant(s), or prior anti-cancer therapy to include: lenalidomide, fludarabine, or alemtuzumab within 12 months; radioimmunoconjugate within 12 weeks; mAb or antibody-drug conjugate within 4 weeks; or radiotherapy/chemotherapy/hormone therapy/targeted small-molecule therapy within 2 weeks prior to Day 1 of Cycle 1
* Active infection
* Positive for human immunodeficiency virus (HIV) or hepatitis B or C
* Receipt of a live virus vaccine within 28 days prior to Day 1 of Cycle 1
* Poor hematologic, renal, or hepatic function
* Pregnant or lactating women
* Life expectancy less than (<) 3 months

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Actual)
Dates: Start 2016-03-24 (Actual); Primary Completion 2021-12-15 (Actual); Study Completion 2021-12-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (28):
- United States (8):
  - Northwest Georgia Oncology Centers, a Service of WellStar Cobb Hospital, Marietta, Georgia
  - Barbara Ann Karmanos Cancer Institute, Detroit, Michigan
  - University of Missouri/Ellis Fischel, Columbia, Missouri
  - Washington University; Wash Uni. Sch. Of Med, St Louis, Missouri
  - NYU School of Medicine, New York, New York
  - Rocky Mountain Cancer Centers, LLP, Irving, Texas
  - Texas Oncology-Tyler, Irving, Texas
  - Texas Oncology San Antonio Medical Center, San Antonio, Texas
- Spain (11):
  - Insititut Catala D'Oncologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital Clínico Málaga, Málaga, Malaga
  - Complejo Hospitalario de Navarra, Pamplona, Navarre
  - Clínica Universidad de Navarra, Pamplona, Navarre
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Clínic. Barcelona, Barcelona
  - Hospital Santa Creu i Sant Pau, Barcelona
  - Hospital Gregorio Marañon, Madrid
  - H. Universitario Leonor, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz., Madrid
  - Hospital La Fe, Valencia
- United Kingdom (9):
  - St James University Hospital, Leeds
  - University Hospitals of Leicester NHS Trust - Leicester Royal Infirmary, Leicester
  - Royal Liverpool University Hospital, Liverpool
  - Barts Hospital; Institute of Cancer, London
  - Sarah Cannon Research Institute, London
  - Maidstone & Tonbridge Wells Hospital; Kent Oncology Center, Maidstone
  - Nottingham University Hospitals NHS Trust - City Hospital, Nottingham
  - Barking, Havering and Redbridge University Hospitals NHS Trust - Queen's Hospital, Romford
  - The Royal Wolverhampton Hospitals NHS Trust; Department of Haematology, Wolverhampton

REFERENCES:
- [Derived] Abrisqueta P, Gonzalez-Barca E, Panizo C, Perez JMA, Miall F, Bastos-Oreiro M, Triguero A, Banerjee L, McMillan A, Seymour E, Hirata J, de Guzman J, Sharma S, Jin HY, Musick L, Diefenbach C. Polatuzumab vedotin plus rituximab and lenalidomide in patients with relapsed or refractory diffuse large B-cell lymphoma: a cohort of a multicentre, single-arm, phase 1b/2 study. Lancet Haematol. 2024 Feb;11(2):e136-e146. doi: 10.1016/S2352-3026(23)00345-9. Epub 2024 Jan 5. PMID 38190832
- [Derived] Diefenbach C, Kahl BS, McMillan A, Briones J, Banerjee L, Cordoba R, Miall F, Burke JM, Hirata J, Jiang Y, Paulson JN, Chang YM, Musick L, Abrisqueta P. Polatuzumab vedotin plus obinutuzumab and lenalidomide in patients with relapsed or refractory follicular lymphoma: a cohort of a multicentre, single-arm, phase 1b/2 study. Lancet Haematol. 2021 Dec;8(12):e891-e901. doi: 10.1016/S2352-3026(21)00311-2. PMID 34826412

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 114 participants with relapsed or refractory (R/R) follicular lymphoma (FL) or diffuse large B-cell lymphoma (DLBCL) were enrolled in this study at 28 investigative sites in Spain, United Kingdom, and United States from 24 March 2016 to 15 December 2021. The study consisted of two phases: dose-escalation and dose-expansion phase. All eligible participants in both phases received induction and post-induction therapy.
Pre-assignment Details: Participants were enrolled in Phase Ib and Phase II study to receive polatuzumab vedotin (pola) in combination with lenalidomide (L) & fixed doses of rituximab (R)/obinutuzumab(G). Of the 114 enrolled participants, 113 participants received at least one dose of the study drug and their intended treatment. One participant withdrew consent prior to receiving any study treatment.
Groups:
- Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL: Participants with FL received lenalidomide, 10 milligrams (mg) capsules orally once daily (QD) on Days 1-21 of Cycles 1 to 6 (1 cycle = 28 days) along with obinutuzumab, 1000 mg, as intravenous (IV) infusion on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of Cycles 2-6, and polatuzumab vedotin, 1.4 milligrams per kilogram (mg/kg), IV infusion on Day 1 of Cycles 1-6, as induction treatment. Thereafter participants who achieved complete response (CR), partial response (PR), or stable disease (SD) at end of induction (EOI) received maintenance treatment until disease progression or unacceptable toxicity for up to 24 months. During maintenance treatment participants received lenalidomide, 10 mg, capsules, orally, QD on Days 1-21 of each month (1 month = 28 days) for up to 12 months, and obinutuzumab, 1000 mg IV on Day 1 of every other month for up to 24 months.
- Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 1000 mg G in FL: Participants with FL received lenalidomide, 10 mg capsules orally QD on Days 1-21 of Cycles 1 to 6 (1 cycle = 28 days) along with obinutuzumab, 1000 mg, as IV infusion on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of Cycles 2-6, and polatuzumab vedotin, 1.8 mg/kg, IV infusion on Day 1 of Cycles 1-6, as induction treatment. Thereafter participants who achieved CR, PR, or SD at EOI received maintenance treatment until disease progression or unacceptable toxicity for up to 24 months. During maintenance treatment participants received lenalidomide, 10 mg, capsules, orally, QD on Days 1-21 of each month (1 month = 28 days) for up to 12 months, and obinutuzumab, 1000 mg IV on Day 1 of every other month for up to 24 months.
- Dose-escalation Phase: 1.4 mg Pola + 15 mg L + 1000 mg G in FL: Participants with FL received lenalidomide, 15 mg capsules orally QD on Days 1-21 of Cycles 1 to 6 (1 cycle = 28 days) along with obinutuzumab, 1000 mg, as IV infusion on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of Cycles 2-6, and polatuzumab vedotin, 1.4 mg/kg, IV infusion on Day 1 of Cycles 1-6, as induction treatment. Thereafter participants who achieved CR, PR, or SD at EOI received maintenance treatment until disease progression or unacceptable toxicity for up to 24 months. During maintenance treatment participants received lenalidomide, 10 mg, capsules, orally, QD on Days 1-21 of each month (1 month = 28 days) for up to 12 months, and obinutuzumab, 1000 mg IV on Day 1 of every other month for up to 24 months.
- Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL; Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL: Participants with FL received lenalidomide, 20 mg capsules orally QD on Days 1-21 of Cycles 1 to 6 (1 cycle = 28 days) along with obinutuzumab, 1000 mg, as IV infusion on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of Cycles 2-6, and polatuzumab vedotin, 1.4 mg/kg, IV infusion on Day 1 of Cycles 1-6, as induction treatment. Thereafter participants who achieved CR, PR, or SD at EOI received maintenance treatment until disease progression or unacceptable toxicity for up to 24 months. During maintenance treatment participants received lenalidomide, 10 mg, capsules, orally, QD on Days 1-21 of each month (1 month = 28 days) for up to 12 months, and obinutuzumab, 1000 mg IV on Day 1 of every other month for up to 24 months.
- Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL: Participants with DLBCL received lenalidomide, 10 mg, capsules orally QD on Days 1-21 of Cycles 1-6 (1 cycle = 28 days) along with rituximab, 375 milligrams per square meter (mg/m^2), as IV infusion on Day 1 of Cycles 1-6 and polatuzumab vedotin, 1.8 mg/kg, as an IV infusion on Day 1 of Cycles 1 to 6, as induction treatment. Thereafter participants who achieved CR or PR at EOI received consolidation treatment until disease progression or unacceptable toxicity for up to 6 months. During consolidation treatment, participants received lenalidomide, 10 mg, capsules, orally, QD on Days 1-21 of each month (1 month = 28 days) for up to 6 months, and rituximab, 375 mg/m^2 IV on Day 1 of every other month for up to 6 months.
- Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL: Participants with DLBCL received lenalidomide, 15 mg, capsules orally QD on Days 1-21 of Cycles 1-6 (1 cycle = 28 days) along with rituximab, 375 mg/m^2, as IV infusion on Day 1 of Cycles 1-6 and polatuzumab vedotin, 1.8 mg/kg, as an IV infusion on Day 1 of Cycles 1 to 6, as induction treatment. Thereafter participants who achieved CR or PR at EOI received consolidation treatment until disease progression or unacceptable toxicity for up to 6 months. During consolidation treatment, participants received lenalidomide, 10 mg, capsules, orally, QD on Days 1-21 of each month (1 month = 28 days) for up to 6 months, and rituximab, 375 mg/m^2 IV on Day 1 of every other month for up to 6 months.
- Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL; Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL: Participants with DLBCL received lenalidomide, 20 mg, capsules orally QD on Days 1-21 of Cycles 1-6 (1 cycle = 28 days) along with rituximab, 375 mg/m^2, as IV infusion on Day 1 of Cycles 1-6 and polatuzumab vedotin, 1.8 mg/kg, as an IV infusion on Day 1 of Cycles 1 to 6, as induction treatment. Thereafter participants who achieved CR or PR at EOI received consolidation treatment until disease progression or unacceptable toxicity for up to 6 months. During consolidation treatment, participants received lenalidomide, 10 mg, capsules, orally, QD on Days 1-21 of each month (1 month = 28 days) for up to 6 months, and rituximab, 375 mg/m^2 IV on Day 1 of every other month for up to 6 months.
Period: Overall Study
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 15 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Started | 3 | 4 | 3 | 6 | 3 | 5 | 10 | 40 | 40
Intent-to-Treat Population (The intent-to-treat (ITT) population included all participants enrolled in the study.) | 3 | 4 | 3 | 6 | 3 | 5 | 10 | 40 | 40
Safety-evaluable Population (The safety-evaluable population included all participants who received at least one dose of any component of the combination.) | 3 | 4 | 3 | 6 | 3 | 5 | 10 | 40 | 39
Immunogenicity-evaluable Population (Immunogenicity population included all safety-evaluable participants with at least one ADA sample.) | 3 | 4 | 3 | 6 | 3 | 5 | 10 | 39 | 38
Pharmacokinetic-evaluable Population (The pharmacokinetic-evaluable population included all participants who received at least one dose of any component of the combination and who provided at least one suitable postdose PK sample.) | 3 | 4 | 3 | 6 | 3 | 5 | 10 | 40 | 39
Completed | 1 | 2 | 2 | 4 | 0 | 3 | 0 | 28 | 17
Not Completed | 2 | 2 | 1 | 2 | 3 | 2 | 10 | 12 | 23
Not completed — Death | 1 | 2 | 1 | 2 | 3 | 2 | 10 | 7 | 20
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 4 | 2
Not completed — Reason Not Specified | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The ITT population included all participants enrolled in the study.
Groups:
- Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL: Participants with FL received lenalidomide, 10 mg capsules orally QD on Days 1-21 of Cycles 1 to 6 (1 cycle = 28 days) along with obinutuzumab, 1000 mg, as IV infusion on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of Cycles 2-6, and polatuzumab vedotin, 1.4 mg/kg, IV infusion on Day 1 of Cycles 1-6, as induction treatment. Thereafter participants who achieved CR, PR, or SD at EOI received maintenance treatment until disease progression or unacceptable toxicity for up to 24 months.
  During maintenance treatment participants received lenalidomide, 10 mg, capsules, orally, QD on Days 1-21 of each month (1 month = 28 days) for up to 12 months, and obinutuzumab, 1000 mg IV on Day 1 of every other month for up to 24 months.
- Total: Total of all reporting groups
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 15 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Total
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 5 | 10 | 40 | 40 | 114
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (6.1) | 72.5 (8.1) | 56.0 (3.5) | 58.3 (12.0) | 59.7 (6.5) | 62.0 (14.9) | 61.4 (14.2) | 61.6 (11.2) | 68.4 (12.8) | 64.0 (12.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 3 | 2 | 4 | 0 | 1 | 4 | 12 | 14 | 42
  Male | 1 | 1 | 1 | 2 | 3 | 4 | 6 | 28 | 26 | 72
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  White | 3 | 4 | 3 | 6 | 3 | 5 | 10 | 36 | 38 | 108
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 1 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Ethnicity: Hispanic or Latino | 0 | 0 | 0 | 0 | 0 | 1 | 3 | 4 | 4 | 12
  Ethnicity: Not Hispanic or Latino | 3 | 4 | 2 | 6 | 3 | 4 | 7 | 34 | 34 | 97
  Ethnicity: Not Stated | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 1 | 4
  Ethnicity: Unknown | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Dose-Limiting Toxicities (DLTs)
Description: A DLT was defined as any one of the following toxicities occurring during the first cycle of treatment and assessed by the investigator as related to study treatment: Any adverse event of any grade that lead to a delay of > 14 days in the start of the next treatment cycle, Grade 3 or 4 non-hematologic adverse events with few exceptions; increase in hepatic transaminase > 3 x baseline and an increase in direct bilirubin > 2 x upper limits of normal (ULN), without any findings of cholestasis or jaundice, or signs of hepatic dysfunction, and in the absence of other contributory factors; hematologic adverse events that met a few protocol specified criteria. DLTs were assessed according to the National Cancer Institute Common Terminology Criteria for Adverse Events, Version 4.0 (NCI CTCAE v4.0). Percentages have been rounded off to the first decimal point.
Time Frame: Day 1 of Cycle 1 to Day 1 of Cycle 2 (1 cycle = 28 days) in dose-escalation phase
Population: The safety-evaluable population included all participants who received at least one dose of any component of the combination.
Measure: Number; unit: percentage of participants
Groups:
- Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL: Participants with DLBCL received lenalidomide, 10 mg, capsules orally QD on Days 1-21 of Cycles 1-6 (1 cycle = 28 days) along with rituximab, 375 milligrams per square meter (mg/m^2), as IV infusion on Day 1 of Cycles 1-6 and polatuzumab vedotin, 1.8 mg/kg, as an IV infusion on Day 1 of Cycles 1 to 6, as induction treatment. Thereafter participants who achieved CR and PR at EOI received consolidation treatment until disease progression or unacceptable toxicity for up to 6 months.
  During consolidation treatment, participants received lenalidomide, 10 mg, capsules, orally, QD on Days 1-21 of each month (1 month = 28 days) for up to 6 months, and rituximab, 375 mg/m^2 IV on Day 1 of every other month for up to 6 months.
- Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL: Participants with DLBCL received lenalidomide, 15 mg, capsules orally QD on Days 1-21 of Cycles 1-6 (1 cycle = 28 days) along with rituximab, 375 mg/m^2, as IV infusion on Day 1 of Cycles 1-6 and polatuzumab vedotin, 1.8 mg/kg, as an IV infusion on Day 1 of Cycles 1 to 6, as induction treatment. Thereafter participants who achieved CR and PR at EOI received consolidation treatment until disease progression or unacceptable toxicity for up to 6 months.
  During consolidation treatment, participants received lenalidomide, 10 mg, capsules, orally, QD on Days 1-21 of each month (1 month = 28 days) for up to 6 months, and rituximab, 375 mg/m^2 IV on Day 1 of every other month for up to 6 months.
- Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL: Participants with DLBCL received lenalidomide, 20 mg, capsules orally QD on Days 1-21 of Cycles 1-6 (1 cycle = 28 days) along with rituximab, 375 mg/m^2, as IV infusion on Day 1 of Cycles 1-6 and polatuzumab vedotin, 1.8 mg/kg, as an IV infusion on Day 1 of Cycles 1 to 6, as induction treatment. Thereafter participants who achieved CR and PR at EOI received consolidation treatment until disease progression or unacceptable toxicity for up to 6 months.
  During consolidation treatment, participants received lenalidomide, 10 mg, capsules, orally, QD on Days 1-21 of each month (1 month = 28 days) for up to 6 months, and rituximab, 375 mg/m^2 IV on Day 1 of every other month for up to 6 months.
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 15 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 5 | 10
percentage of participants | 0.0 | 50.0 | 0.0 | 0.0 | 0.0 | 0.0 | 0.0

2. Primary Outcome: Percentage of Participants With Adverse Events (AEs)
Description: An AE is any untoward medical occurrence in a participant administered a pharmaceutical product and which does not necessarily have to have a causal relationship with the treatment. An AE can therefore be any unfavorable and unintended sign (including an abnormal laboratory finding, for example), symptom, or disease temporally associated with the use of a pharmaceutical product, whether or not considered related to the pharmaceutical product. Preexisting conditions which worsen during a study are also considered as adverse events. Percentages have been rounded off to the first decimal point.
Time Frame: From study start up to end of study (Up to a maximum of 69 months)
Population: as for outcome 1
Measure: Number; unit: percentage of participants
Groups:
- Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL: Participants with DLBCL received lenalidomide, 20 mg, capsules orally QD on Days 1-21 of Cycles 1-6 (1 cycle = 28 days) along with rituximab, 375 mg/m^2, as IV infusion on Day 1 of Cycles 1-6 and polatuzumab vedotin, 1.8 mg/kg, as an IV infusion on Day 1 of Cycles 1 to 6, as induction treatment. Thereafter participants who achieved CR and PR at EOI received consolidation treatment until disease progression or unacceptable toxicity for up to 6 months.
  During consolidation treatment, participants received lenalidomide, 10 mg, capsules, orally, QD on Days 1-21 of each month (1 month = 28 days) for up to 6 months, and rituximab, 375 mg/m^2 IV on Day 1 of every other month for up to 6 months.
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 15 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 5 | 10 | 40 | 39
percentage of participants | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 100.0 | 97.4

3. Primary Outcome: Percentage of Participants With Complete Response (CR) at End of Induction (EOI), Determined by an Independent Review Committee (IRC) on the Basis of Positron Emission Tomography (PET) and Computed Tomography (CT) Scans
Description: CR at EOI was assessed by IRC according to Modified Lugano Response Criteria (MLRC). Per MLRC, CR based on PET-CT was defined as complete metabolic response (MR) in lymph nodes and extralymphatic sites (ELS) with a score of 1, 2, or 3 with or without residual mass, on 5-point scale (5PS) where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake > mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions no evidence of fluorodeoxyglucose (FDG)-avid disease in bone marrow. Bone marrow is normal by morphology; if indeterminate, immunohistochemistry (IHC) negative. Analysis was done 6-8 weeks after Cycle 6, Day 1 (cycle=28 days). Percentages have been rounded off to the first decimal point.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks)
Population: Efficacy-evaluable population=dose expansion participants who received atleast 1 dose of any component of the combination. As pre-specified in the protocol, data was collected and analysed only for participants in expansion phase arms & those participants in dose-escalation arms who received study drugs at RP2D (i.e. arms: 1.4 mg Pola + 20 mg L+1000G for FL; 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL), for this OM.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 6 | 10 | 40 | 39
percentage of participants | 66.7 [27.13 to 93.72] | 0.0 [0.0 to 25.89] | 60.0 [45.78 to 73.06] | 38.5 [25.41 to 52.89]

4. Secondary Outcome: Percentage of Participants With CR at EOI, Determined by the Investigator on the Basis of PET-CT Scans
Description: CR at EOI was assessed by Investigator according to MLRC. Per MLRC, CR based on PET-CT was defined as complete MR in lymph nodes and ELS with a score of 1, 2, or 3 with or without residual mass, on 5PS where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake > mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions no evidence of FDG-avid disease in bone marrow. Bone marrow is normal by morphology; if indeterminate, IHC negative. Analysis was done 6-8 weeks after Cycle 6, Day 1 (cycle=28 days). Percentages have been rounded off to the first decimal point.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 6 | 10 | 40 | 39
percentage of participants | 66.7 [27.13 to 93.72] | 0.0 [0.0 to 25.89] | 60.0 [45.78 to 73.06] | 33.3 [20.97 to 47.69]

5. Secondary Outcome: Percentage of Participants With CR at EOI, Determined by the IRC on the Basis of CT Scans Alone
Description: CR at EOI was determined by IRC according to the MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in longest transverse diameter (LDi) and no ELS of disease organ enlargement regressing to normal; no new lesions; normal bone marrow by morphology, if indeterminate, IHC negative. Analysis was done 6-8 weeks after Cycle 6, Day 1 (cycle=28 days). Percentages have been rounded off to the first decimal point.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks)
Population: Efficacy-evaluable population=dose expansion participants who received atleast 1 dose of any component of the combination. As pre-specified in the protocol, data was collected and analysed only for participants in expansion phase arms & those participants in dose-escalation arms who received study drugs at RP2D (i.e. arms: 1.4 mg Pola + 20 mg L+1000G for FL; 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL), for this OM. 'Overall Number Analyzed'=number of participants with data available for analysis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Groups:
- Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL: Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL Participants with FL received lenalidomide, 20 mg capsules orally QD on Days 1-21 of Cycles 1 to 6 (1 cycle = 28 days) along with obinutuzumab, 1000 mg, as IV infusion on Days 1, 8, and 15 of Cycle 1 and then on Day 1 of Cycles 2-6, and polatuzumab vedotin, 1.4 mg/kg, IV infusion on Day 1 of Cycles 1-6, as induction treatment. Thereafter participants who achieved CR, PR, or SD at EOI received maintenance treatment until disease progression or unacceptable toxicity for up to 24 months. During maintenance treatment participants received lenalidomide, 10 mg, capsules, orally, QD on Days 1-21 of each month (1 month = 28 days) for up to 12 months, and obinutuzumab, 1000 mg IV on Day 1 of every other month for up to 24 months.
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 6 | 8 | 35 | 32
percentage of participants | 16.7 [0.85 to 58.18] | 0.0 [0.0 to 31.23] | 31.4 [18.73 to 46.61] | 12.5 [4.38 to 26.36]

6. Secondary Outcome: Percentage of Participants With CR at EOI, Determined by Investigator on the Basis of CT Scans Alone
Description: CR at EOI was determined by Investigator according to the MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no ELS of disease organ enlargement regressing to normal; no new lesions; normal bone marrow by morphology, if indeterminate, IHC negative. Analysis was done 6-8 weeks after Cycle 6, Day 1 (cycle=28 days). Percentages have been rounded off to the first decimal point.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks)
Population: as for outcome 5
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 6 | 9 | 37 | 32
percentage of participants | 16.7 [0.85 to 58.18] | 0.0 [0.0 to 28.31] | 29.7 [17.65 to 44.38] | 28.1 [15.53 to 43.94]

7. Secondary Outcome: Percentage of Participants With Objective Response (OR) at EOI, Determined by the IRC on the Basis of PET-CT Scans
Description: OR was defined as percentage of participants with CR or PR as assessed by the IRC according to MLRC. Per MLRC CR based on PET-CT is complete MR in lymph nodes & ELS with score of 1, 2, or 3 with or without residual mass on 5PS, where 1=no uptake above background; 2=uptake ≤ mediastinum; 3=uptake> mediastinum but ≤ liver; 4=uptake moderately > liver; 5=uptake markedly higher than liver and/or new lesions;no new lesions & no evidence of FDG-avid disease in bone marrow.Bone marrow is normal by morphology; if indeterminate, IHC negative. Partial response (PR) based on PET-CT was defined as partial MR in lymph nodes & ELS with score of 4 or 5 with reduced uptake compared with baseline & residual masses of any size at interim, residual uptake higher than uptake in normal bone marrow but reduced compared with baseline (diffuse uptake compatible with reactive changes from chemotherapy allowed). Percentages have been rounded off up to the second decimal point.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (cycle=28 days) (up to approximately 28 weeks)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 6 | 10 | 40 | 39
percentage of participants | 100.0 [60.70 to 100.0] | 10.0 [0.51 to 39.42] | 72.50 [58.61 to 83.75] | 46.20 [32.35 to 60.42]

8. Secondary Outcome: Percentage of Participants With Objective Response at EOI, Determined by Investigator on the Basis of PET-CT Scans
Description: OR was defined percentage of participants with CR or PR assessed by the investigator according to MLRC. Per MLRC CR based on PET-CT is complete MR in lymph nodes & ELS with score of 1, 2, 3 with or without residual mass on 5PS, where 1=no uptake above background 2=uptake ≤ mediastinum 3=uptake> mediastinum but ≤ liver 4=uptake moderately > liver 5=uptake markedly higher than liver and/or new lesions;no new lesions & no evidence of FDG-avid disease in bone marrow.Bone marrow is normal by morphology; if indeterminate, IHC negative. PR based on PET-CT was defined as partial MR in lymph nodes & ELS with score of 4 or 5 with reduced uptake compared with baseline & residual masses of any size at interim, residual uptake higher than uptake in normal bone marrow but reduced compared with baseline(diffuse uptake compatible with reactive changes from chemotherapy allowed). Percentages are rounded off.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 6 | 10 | 40 | 39
percentage of participants | 100.0 [60.70 to 100.0] | 10.0 [0.51 to 39.42] | 80.0 [66.80 to 89.64] | 46.20 [32.35 to 60.42]

9. Secondary Outcome: Percentage of Participants With Objective Response at EOI, Determined by the IRC on the Basis of CT Scans Alone
Description: OR was defined as the percentage of participants with CR or PR, as assessed by the IRC based on MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no ELS of disease organ enlargement regressing to normal; no new lesions; bone marrow normal by morphology, if indeterminate, IHC negative. PR per CT only was defined as partial remission in lymph nodes and ELS with ≥50% decrease in the sum of the products of greatest diameters (SPD) of up to 6 target measurable lymph nodes and extranodal sites, absent/normal/regressed but with no increase in non-measured lesions, spleen regressing by ≥50% in length beyond normal it, no new sites of lesions. The analysis was done 6-8 weeks after Cycle 6, Day 1 (each cycle is 28 days). Percentages have been rounded off to the first decimal point.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks)
Population: as for outcome 5
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 6 | 8 | 35 | 32
percentage of participants | 100.0 [60.70 to 100.0] | 12.5 [0.64 to 47.07] | 91.4 [79.31 to 97.62] | 53.1 [37.34 to 68.46]

10. Secondary Outcome: Percentage of Participants With Objective Response, Determined by the Investigator on the Basis of CT Scans Alone
Description: OR was defined as the percentage of participants with CR or PR, as assessed by the investigator based on MLRC. Per MLRC, CR based on CT was defined as complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no ELS of disease organ enlargement regressing to normal; no new lesions; bone marrow normal by morphology, if indeterminate, IHC negative. PR per CT only was defined as partial remission in lymph nodes and ELS with ≥50% decrease in the sum of the products of greatest diameters (SPD) of up to 6 target measurable lymph nodes and extranodal sites, absent/normal/regressed but with no increase in non-measured lesions, spleen regressing by ≥50% in length beyond normal it, no new sites of lesions. Analysis was done 6-8 weeks after Cycle 6, Day 1 (cycle=28 days). Percentages have been rounded off to the first decimal point.
Time Frame: 6 to 8 weeks after Day 1 of Cycle 6 (up to approximately 28 weeks)
Population: as for outcome 5
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 6 | 9 | 37 | 32
percentage of participants | 100.0 [60.70 to 100.0] | 11.1 [0.57 to 42.91] | 89.2 [76.95 to 96.22] | 59.4 [43.35 to 74.03]

11. Secondary Outcome: Percentage of Participants With Best Response of CR or PR, Determined by the Investigator on the Basis of CT Scans Alone
Description: BOR=CR/PR per CT per MLRC. Per MLRC, CR based on CT was defined as a complete radiologic response in lymph nodes and ELS with target nodes/nodal masses regressing to ≤ 1.5 cm in LDi and no ELS of disease organ enlargement regressing to normal; no new lesions; bone marrow normal by morphology, if indeterminate, IHC negative. PR per CT only was defined as partial remission in lymph nodes and ELS with ≥50% decrease in SPD of up to 6 target measurable lymph nodes and extranodal sites, absent/normal/regressed but with no increase in non-measured lesions, spleen regressing by ≥50% in length beyond normal it, no new sites of lesions. Percentages have been rounded off to the first decimal point.
Time Frame: Up to every 6 months until disease progression, unacceptable toxicity or study completion (up to approximately 69 months)
Population: as for outcome 3
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 6 | 10 | 40 | 39
percentage of participants | 100.0 [60.70 to 100.0] | 50.0 [22.24 to 77.76] | 90.0 [78.56 to 96.51] | 79.5 [66.02 to 89.36]

12. Secondary Outcome: Observed Serum Obinutuzumab Concentration
Description: 1 cycle = 28 days
Time Frame: Day 1 of Cycles 1, 2, 4 & 6: predose & 30 mins postdose; EOI: predose; Day 1 of Maintenance Months 1,7, 13, 19;Day 120 post last dose; one year post last dose; study drug discontinuation; unscheduled visit: predose (up to approximately 69 months)
Population: The pharmacokinetic (PK)-evaluable population included all participants who received at least one dose of any component of the combination and who provided at least one suitable postdose PK sample. 'Overall Number Analyzed' is the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: micrograms per milliliter (μg/mL)
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 15 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 38
micrograms per milliliter (μg/mL)
  Induction Cycle 1 Day 1 / Predose: number analyzed (Participants) | 3 | 4 | 2 | 6 | 37
  Induction Cycle 1 Day 1 / Predose | NA (NA) — The data is not evaluable as the samples were below lower limit of quantification (BLLQ). | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ.
  Induction Cycle 1 Day 1 / 30 mins: number analyzed (Participants) | 3 | 3 | 3 | 4 | 35
  Induction Cycle 1 Day 1 / 30 mins | 394 (22.1) | 358 (20.5) | 351 (15.2) | 333 (70.0) | 182 (206.7)
  Induction Cycle 2 Day 1 / Predose: number analyzed (Participants) | 3 | 3 | 3 | 4 | 36
  Induction Cycle 2 Day 1 / Predose | 451 (23.5) | 372 (37.0) | 386 (4.6) | 481 (23.1) | 312 (40.8)
  Induction Cycle 2 Day 1 / 30 mins: number analyzed (Participants) | 3 | 3 | 3 | 5 | 36
  Induction Cycle 2 Day 1 / 30 mins | 830 (38.3) | 749 (17.2) | 695 (14.3) | 667 (77.5) | 588 (41.4)
  Induction Cycle 4 Day 1 / Predose: number analyzed (Participants) | 3 | 2 | 2 | 4 | 34
  Induction Cycle 4 Day 1 / Predose | 354 (15.0) | 321 (43.6) | 344 (13.4) | 405 (24.9) | 270 (41.8)
  Induction Cycle 4 Day 1 / 30 mins: number analyzed (Participants) | 1 | 2 | 2 | 5 | 33
  Induction Cycle 4 Day 1 / 30 mins | 103 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 644 (42.8) | 653 (20.6) | 742 (27.8) | 547 (37.1)
  Induction Cycle 6 Day 1 / Predose: number analyzed (Participants) | 3 | 1 | 2 | 5 | 34
  Induction Cycle 6 Day 1 / Predose | 255 (36.6) | 504 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 327 (5.8) | 384 (52.2) | 255 (49.0)
  Induction Cycle 6 Day 1 / 30 mins: number analyzed (Participants) | 3 | 1 | 2 | 5 | 33
  Induction Cycle 6 Day 1 / 30 mins | 730 (15.5) | 804 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 1.18 (NA) — Values were less than reportable (LTR) for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not calculated. | 751 (35.3) | 543 (36.2)
  EOI / Predose: number analyzed (Participants) | 3 | 0 | 0 | 0 | 0
  EOI / Predose | 108 (32.6) |  |  |  |
  Maintenance Month 1 / Predose: number analyzed (Participants) | 2 | 1 | 0 | 4 | 27
  Maintenance Month 1 / Predose | 231 (19.1) | 381 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 230 (87.4) | 176 (60.1)
  Maintenance Month 7 / Predose: number analyzed (Participants) | 1 | 1 | 1 | 3 | 21
  Maintenance Month 7 / Predose | 128 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 212 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 229 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 125 (143.7) | 135 (64.3)
  Maintenance Month 13 / Predose: number analyzed (Participants) | 0 | 1 | 1 | 3 | 18
  Maintenance Month 13 / Predose |  | 142 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 269 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 134 (105.3) | 150 (70.7)
  Maintenance Month 19 / Predose: number analyzed (Participants) | 0 | 1 | 1 | 2 | 15
  Maintenance Month 19 / Predose |  | 354 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 204 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 154 (144.1) | 165 (59.5)
  Study Drug Discontinuation: number analyzed (Participants) | 0 | 1 | 0 | 1 | 10
  Study Drug Discontinuation |  | 46.4 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 17.3 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 87.5 (588.7)
  Day 120 Post Last Dose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 7
  Day 120 Post Last Dose | 29.1 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  |  |  | 44.5 (806.5)
  1 Year Post Last Dose: number analyzed (Participants) | 0 | 0 | 1 | 0 | 7
  1 Year Post Last Dose |  |  | 0.377 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 0.340 (955.9)
  Unscheduled / Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 1
  Unscheduled / Predose |  |  |  |  | 561 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated.

13. Secondary Outcome: Observed Serum Rituximab Concentration
Time Frame: Day 1 of Cycles 1, 2, 4, 6: predose and 30 mins post-dose (1 cycle = 28 days) (up to approximately 69 months)
Population: The PK-evaluable population included all participants who received at least one dose of any component of the combination and who provided at least one suitable PK samples. 'Overall Number Analyzed' is the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoint.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 3 | 5 | 10 | 37
μg/mL
  Induction Cycle 1 Day 1 / Predose: number analyzed (Participants) | 2 | 5 | 10 | 36
  Induction Cycle 1 Day 1 / Predose | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ.
  Induction Cycle 1 Day 1 / 30 mins: number analyzed (Participants) | 2 | 4 | 9 | 36
  Induction Cycle 1 Day 1 / 30 mins | 151 (42.9) | 203 (28.1) | 175 (18.7) | 174 (45.4)
  Induction Cycle 2 Day 1 / Predose: number analyzed (Participants) | 3 | 3 | 7 | 34
  Induction Cycle 2 Day 1 / Predose | 25.6 (78.0) | 33.3 (43.7) | 31.7 (26.2) | 26.4 (73.4)
  Induction Cycle 2 Day 1 / 30 mins: number analyzed (Participants) | 1 | 1 | 1 | 32
  Induction Cycle 2 Day 1 / 30 mins | 133 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 172 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 222 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 194 (36.4)
  Induction Cycle 4 Day 1 / Predose: number analyzed (Participants) | 1 | 2 | 4 | 27
  Induction Cycle 4 Day 1 / Predose | 20.4 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 74.6 (33.8) | 53.1 (43.7) | 58.3 (44.4)
  Induction Cycle 4 Day 1 / 30 mins: number analyzed (Participants) | 1 | 2 | 4 | 26
  Induction Cycle 4 Day 1 / 30 mins | 159 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 224 (5.7) | 220 (16.2) | 228 (36.6)
  Induction Cycle 6 Day 1 / Predose: number analyzed (Participants) | 1 | 3 | 2 | 19
  Induction Cycle 6 Day 1 / Predose | 15.3 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 79.5 (42.3) | 74.7 (22.1) | 68.9 (60.6)
  Induction Cycle 6 Day 1 / 30 mins: number analyzed (Participants) | 1 | 2 | 2 | 19
  Induction Cycle 6 Day 1 / 30 mins | 135 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 250 (7.6) | 233 (1.8) | 256 (26.4)

14. Secondary Outcome: Serum Concentration of Polatuzumab Vedotin Analyte: Total Antibody
Time Frame: Day 1 of Cycles 1, 2, 4: predose (1 cycle = 28 days), Day 120 post last dose; one year post last dose; study drug discontinuation; unscheduled visit: predose (up to approximately 69 months)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 15 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 4 | 7 | 37 | 37
μg/mL
  Induction Cycle 1 Day 1 / Predose: number analyzed (Participants) | 3 | 4 | 2 | 6 | 3 | 4 | 7 | 36 | 37
  Induction Cycle 1 Day 1 / Predose | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ.
  Induction Cycle 2 Day 1 / Predose: number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 7 | 37 | 35
  Induction Cycle 2 Day 1 / Predose | 1.47 (16.2) | 2.01 (51.1) | 0.200 (958.3) | 0.622 (152.8) | 1.57 (62.9) | 1.61 (59.8) | 1.47 (26.2) | 0.339 (391.8) | 1.35 (122.0)
  Induction Cycle 4 Day 1 / Predose: number analyzed (Participants) | 3 | 2 | 2 | 5 | 1 | 3 | 4 | 35 | 26
  Induction Cycle 4 Day 1 / Predose | 1.83 (51.7) | 4.45 (20.5) | 2.57 (30.5) | 2.12 (69.0) | 0.900 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 2.96 (44.4) | 3.10 (43.6) | 2.31 (48.5) | 3.42 (46.1)
  Study Drug Discontinuation: number analyzed (Participants) | 3 | 1 | 0 | 2 | 1 | 1 | 3 | 11 | 18
  Study Drug Discontinuation | 0.106 (209.1) | 0.170 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 0.0903 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not calculated. | 1.50 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 6.16 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 3.25 (49.7) | 0.175 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated. | 0.455 (448.4)
  Day 120 Post Last Dose: number analyzed (Participants) | 1 | 0 | 0 | 0 | 0 | 1 | 1 | 9 | 9
  Day 120 Post Last Dose | 0.0661 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  |  |  |  | 0.208 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 0.107 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 0.0365 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated. | 0.0666 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated.
  1 Year Post Last Dose: number analyzed (Participants) | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 7 | 9
  1 Year Post Last Dose | 0.0250 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 0.0250 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  |  |  |  | 0.0357 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated. | 0.0250 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated.
  Unscheduled / Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
  Unscheduled / Predose |  |  |  |  |  |  |  |  | 2.59 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated.

15. Secondary Outcome: Plasma Concentration of Polatuzumab Vedotin Analyte: Antibody-conjugated MMAE (acMMAE)
Time Frame: Day 1 of Cycles 1, 2, 4: predose and 30 mins post-dose; Days 8 and 15 of Cycle 1; Day 1 of Cycle 6: predose, study drug discontinuation; unscheduled visit: predose (1 cycle = 28 days) (up to approximately 69 months)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: nanograms per milliliter (ng/mL)
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 15 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 5 | 10 | 40 | 39
nanograms per milliliter (ng/mL)
  Induction Cycle 1 Day 1 / Predose: number analyzed (Participants) | 3 | 4 | 2 | 6 | 3 | 5 | 10 | 38 | 38
  Induction Cycle 1 Day 1 / Predose | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ.
  Induction Cycle 1 Day 1 / 30 mins: number analyzed (Participants) | 2 | 4 | 3 | 6 | 3 | 5 | 10 | 34 | 36
  Induction Cycle 1 Day 1 / 30 mins | 580 (41.6) | 660 (24.7) | 476 (16.0) | 432 (27.9) | 568 (27.7) | 106 (60902.6) | 513 (73.5) | 333 (267.2) | 522 (323.0)
  Induction Cycle 1 Day 8: number analyzed (Participants) | 3 | 3 | 3 | 5 | 3 | 5 | 7 | 35 | 36
  Induction Cycle 1 Day 8 | 50.2 (7.3) | 80.0 (17.6) | 11.4 (232.2) | 27.7 (69.2) | 58.9 (44.4) | 52.0 (36.3) | 43.9 (96.4) | 11.9 (799.0) | 56.6 (90.2)
  Induction Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 5 | 2 | 5 | 7 | 33 | 33
  Induction Cycle 1 Day 15 | 17.3 (5.5) | 24.7 (13.8) | 2.50 (483.1) | 6.73 (118.8) | 22.3 (31.2) | 18.3 (48.7) | 18.6 (30.5) | 5.95 (366.1) | 16.9 (118.6)
  Induction Cycle 2 Day 1 / Predose: number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 7 | 38 | 33
  Induction Cycle 2 Day 1 / Predose | 4.96 (21.3) | 6.55 (58.7) | 0.961 (477.5) | 2.50 (119.8) | 7.44 (40.2) | 5.58 (77.2) | 6.12 (18.1) | 1.88 (490.2) | 5.32 (103.6)
  Induction Cycle 2 Day 1 / 30 mins: number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 7 | 36 | 31
  Induction Cycle 2 Day 1 / 30 mins | 555 (15.8) | 623 (18.4) | 508 (22.7) | 295 (174.6) | 537 (40.3) | 568 (14.1) | 716 (16.5) | 481 (54.3) | 451 (391.7)
  Induction Cycle 4 Day 1 / Predose: number analyzed (Participants) | 3 | 1 | 2 | 5 | 1 | 3 | 4 | 36 | 26
  Induction Cycle 4 Day 1 / Predose | 5.34 (73.9) | 11.5 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 8.47 (19.5) | 7.68 (60.8) | 4.19 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 8.25 (59.4) | 11.7 (74.2) | 8.99 (36.7) | 11.3 (45.2)
  Induction Cycle 4 Day 1 / 30 mins: number analyzed (Participants) | 2 | 2 | 2 | 5 | 1 | 3 | 4 | 34 | 24
  Induction Cycle 4 Day 1 / 30 mins | 32.9 (101980.7) | 416 (87.7) | 519 (9.3) | 531 (17.6) | 371 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 507 (42.8) | 737 (20.8) | 492 (22.3) | 645 (107.2)
  Induction Cycle 6 Day 1 / Predose: number analyzed (Participants) | 3 | 1 | 2 | 5 | 1 | 3 | 2 | 33 | 21
  Induction Cycle 6 Day 1 / Predose | 7.70 (26.0) | 19.9 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 9.37 (42.6) | 9.70 (53.0) | 3.06 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 11.5 (41.6) | 15.8 (45.4) | 9.82 (40.4) | 11.8 (66.0)
  Study Drug Discontinuation: number analyzed (Participants) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 0
  Study Drug Discontinuation | 0.180 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not calculated. | 0.635 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 0.180 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  |  |  | 1.71 (378.4) |
  Unscheduled / Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1
  Unscheduled / Predose |  |  |  |  |  |  |  | 23.1 (62.5) | 9.78 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated.

16. Secondary Outcome: Plasma Concentration of Polatuzumab Vedotin Analyte: Unconjugated MMAE
Time Frame: Day 1 of Cycles 1, 2, 4: predose and 30 mins post-dose; Days 8 and 15 of Cycle 1 and Day 1 of Cycle 6: predose, study drug discontinuation; unscheduled visit: predose (1 cycle = 28 days) (up to approximately 69 months)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 15 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 5 | 10 | 40 | 39
ng/mL
  Induction Cycle 1 Day 1 / Predose: number analyzed (Participants) | 3 | 4 | 2 | 6 | 3 | 5 | 10 | 38 | 38
  Induction Cycle 1 Day 1 / Predose | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ.
  Induction Cycle 1 Day 1 / 30 mins: number analyzed (Participants) | 2 | 4 | 3 | 6 | 3 | 5 | 10 | 35 | 36
  Induction Cycle 1 Day 1 / 30 mins | 0.228 (7.8) | 0.160 (69.9) | 0.420 (100.6) | 0.233 (74.0) | 0.156 (62.1) | 0.167 (214.8) | 0.298 (198.7) | 0.347 (327.5) | 0.297 (111.1)
  Induction Cycle 1 Day 8: number analyzed (Participants) | 3 | 4 | 3 | 5 | 3 | 5 | 7 | 37 | 36
  Induction Cycle 1 Day 8 | 1.15 (34.9) | 2.05 (49.7) | 2.40 (102.0) | 1.64 (135.5) | 1.89 (76.1) | 1.36 (29.6) | 3.65 (75.3) | 1.12 (227.0) | 2.56 (144.8)
  Induction Cycle 1 Day 15: number analyzed (Participants) | 3 | 3 | 3 | 6 | 2 | 5 | 7 | 33 | 34
  Induction Cycle 1 Day 15 | 0.457 (56.3) | 0.459 (54.5) | 0.387 (6.0) | 0.435 (129.5) | 0.485 (204.0) | 0.456 (39.8) | 0.683 (63.3) | 0.294 (170.9) | 0.843 (125.2)
  Induction Cycle 2 Day 1 / Predose: number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 7 | 38 | 34
  Induction Cycle 2 Day 1 / Predose | 0.0280 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated. | 0.0315 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated. | 0.0244 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated. | 0.0334 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated. | 0.0501 (149.0) | 0.0310 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated. | 0.0527 (102.8) | 0.0268 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated. | 0.0713 (125.0)
  Induction Cycle 2 Day 1 / 30 mins: number analyzed (Participants) | 3 | 3 | 3 | 6 | 3 | 3 | 7 | 36 | 31
  Induction Cycle 2 Day 1 / 30 mins | 0.151 (68.6) | 0.138 (133.0) | 0.151 (49.8) | 0.136 (339.9) | 0.186 (51.2) | 0.123 (53.8) | 0.157 (72.5) | 0.102 (101.2) | 0.210 (77.3)
  Induction Cycle 4 Day 1 / Predose: number analyzed (Participants) | 3 | 1 | 2 | 5 | 1 | 3 | 4 | 36 | 26
  Induction Cycle 4 Day 1 / Predose | 0.0431 (NA) — Values were LTR for 2 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not calculated. | 0.117 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 0.0672 (56.9) | 0.0283 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated. | 0.0180 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 0.0344 (61.0) | 0.0729 (11.4) | 0.0366 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated. | 0.0776 (101.5)
  Induction Cycle 4 Day 1 / 30 mins: number analyzed (Participants) | 2 | 2 | 2 | 5 | 1 | 3 | 4 | 34 | 39
  Induction Cycle 4 Day 1 / 30 mins | 0.0817 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not calculated. | 0.156 (18.7) | 0.104 (7.1) | 0.0752 (113.2) | 0.0180 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 0.133 (50.9) | 0.208 (44.9) | 0.102 (57.7) | 0.213 (51.3)
  Induction Cycle 6 Day 1 / Predose: number analyzed (Participants) | 3 | 1 | 2 | 5 | 1 | 3 | 2 | 33 | 21
  Induction Cycle 6 Day 1 / Predose | 0.0367 (68.3) | 0.0929 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 0.0821 (93.8) | 0.0267 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated. | 0.0180 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 0.0517 (118.9) | 0.0405 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not calculated. | 0.0342 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated. | 0.0852 (62.6)
  Study Drug Discontinuation: number analyzed (Participants) | 2 | 1 | 0 | 1 | 0 | 0 | 0 | 4 | 0
  Study Drug Discontinuation | 0.0180 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not calculated. | 0.0180 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  | 0.0180 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. |  |  |  | 0.0180 (NA) — Since more than one-third values were less than reportable, the geometric coefficient of variation was not calculated. |
  Unscheduled / Predose: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Unscheduled / Predose |  |  |  |  |  |  |  | 0.180 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 0.0180 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated.

17. Secondary Outcome: Observed Plasma Lenalidomide Concentration
Time Frame: Day 1 Cycle 1: predose and 2 hours (hr) post-dose; Day 15 Cycle 1: predose, 0.5hr, 1hr, 2hr, 4hr, 8hr post-dose; Day 1 Cycle 6: 2hr post-dose; unscheduled visits: 2hr post-dose (1 cycle = 28 days) (up to approximately 69 months)
Population: as for outcome 13
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 15 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 4 | 10 | 37 | 37
ng/mL
  Induction Cycle 1 Day 1 / Predose: number analyzed (Participants) | 3 | 4 | 2 | 5 | 3 | 4 | 9 | 36 | 36
  Induction Cycle 1 Day 1 / Predose | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ. | NA (NA) — The data is not evaluable as the samples were BLLQ.
  Induction Cycle 1 Day 1 / 2h: number analyzed (Participants) | 3 | 4 | 3 | 5 | 3 | 4 | 10 | 37 | 36
  Induction Cycle 1 Day 1 / 2h | 118 (44.0) | 144 (30.3) | 201 (54.0) | 305 (37.1) | 25.2 (239.4) | 237 (47.4) | 197 (184.1) | 306 (43.1) | 277 (60.0)
  Induction Cycle 1 Day 15 / Predose: number analyzed (Participants) | 3 | 3 | 2 | 6 | 2 | 4 | 7 | 32 | 31
  Induction Cycle 1 Day 15 / Predose | 5.97 (628.0) | 0.729 (540.0) | 8.74 (277.0) | 5.20 (275.1) | 5.43 (9.1) | 2.64 (68.0) | 8.33 (112.0) | 9.99 (260.9) | 10.4 (196.4)
  Induction Cycle 1 Day 15 / 30 min: number analyzed (Participants) | 3 | 2 | 2 | 4 | 2 | 3 | 7 | 30 | 30
  Induction Cycle 1 Day 15 / 30 min | 64.0 (1553.1) | 1.95 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not calculated. | 179 (220.1) | 202 (115.6) | 12.5 (76.4) | 41.7 (546.7) | 73.3 (395.5) | 124 (300.3) | 94.5 (204.9)
  Induction Cycle 1 Day 15 / 1h: number analyzed (Participants) | 3 | 3 | 2 | 5 | 2 | 3 | 7 | 33 | 30
  Induction Cycle 1 Day 15 / 1h | 61.4 (1354.8) | 40.8 (183.1) | 189 (48.0) | 272 (48.2) | 69.9 (10.3) | 224 (76.8) | 187 (150.5) | 236 (147.7) | 245 (106.8)
  Induction Cycle 1 Day 15 / 2h: number analyzed (Participants) | 3 | 3 | 2 | 5 | 2 | 3 | 7 | 32 | 31
  Induction Cycle 1 Day 15 / 2h | 117 (53.2) | 93.3 (40.5) | 202 (36.0) | 200 (45.5) | 118 (22.3) | 232 (25.5) | 328 (38.2) | 305 (53.6) | 242 (297.2)
  Induction Cycle 1 Day 15 / 4h: number analyzed (Participants) | 3 | 3 | 2 | 4 | 2 | 3 | 7 | 33 | 31
  Induction Cycle 1 Day 15 / 4h | 96.4 (62.0) | 65.7 (46.3) | 116 (28.9) | 152 (36.9) | 79.9 (28.2) | 134 (23.6) | 245 (36.3) | 214 (41.1) | 205 (45.4)
  Induction Cycle 1 Day 15 / 8h: number analyzed (Participants) | 3 | 3 | 2 | 5 | 2 | 3 | 7 | 28 | 30
  Induction Cycle 1 Day 15 / 8h | 35.0 (109.1) | 29.2 (55.2) | 56.8 (57.2) | 49.8 (23.3) | 44.0 (40.2) | 57.0 (19.1) | 105 (50.9) | 103 (56.3) | 103 (67.6)
  Induction Cycle 6 Day 1 / 2h: number analyzed (Participants) | 3 | 1 | 2 | 5 | 2 | 3 | 2 | 33 | 19
  Induction Cycle 6 Day 1 / 2h | 124 (21.4) | 76.1 (NA) — Since only 1 participant was analyzed, the geometric coefficient of variation was not calculated. | 110 (35.1) | 227 (48.1) | 36.2 (NA) — Values were LTR for 1 participant. Since data was evaluable only for 1 participant geometric co-efficient of variation was not calculated. | 258 (10.5) | 255 (36.5) | 237 (52.1) | 153 (515.5)
  Unscheduled / 2h: number analyzed (Participants) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 0
  Unscheduled / 2h |  |  |  |  |  |  |  | 199 (53.3) |

18. Secondary Outcome: Number of Participants With Human Anti-human Antibodies (HAHAs) to Obinutuzumab
Description: The number of participants with positive results for HAHAs, also called anti-drug antibodies (ADAs) against obinutuzumab at baseline and at any of the post-baseline assessment time-points were reported. Number of participants positive for Treatment Emergent ADA = the number of post-baseline evaluable participants determined to have treatment induced ADA or treatment-enhanced ADA during the study period. Treatment-induced ADA = negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result. Treatment-enhanced ADA = a participant with positive ADA result at baseline who has one or more post-baseline titer results that are at least 0.60 titer unit (t.u.) greater than the baseline titer result.
Time Frame: Baseline up to approximately 2 years after last dose (up to approximately 69 months)
Population: Immunogenicity population included all safety-evaluable participants with at least one ADA Sample. 'Overall Number Analyzed' is the number of participants with data available for analysis. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 15 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL
Number analyzed (Participants) | 3 | 4 | 2 | 6 | 38
Participants
  Baseline prevalence of ADAs | 0 | 0 | 0 | 0 | 3
  Post baseline incidence of ADAs: number analyzed (Participants) | 3 | 2 | 2 | 6 | 36
  Post baseline incidence of ADAs | 0 | 0 | 0 | 0 | 0

19. Secondary Outcome: Number of Participants With Human Anti-chimeric Antibodies (HACAs) to Rituximab
Description: The number of participants with positive results for HACAs, also called ADAs against rituximab at baseline and at any of the post-baseline assessment time-points were reported. Number of participants positive for Treatment Emergent ADA = the number of post-baseline evaluable participants determined to have treatment induced ADA or treatment-enhanced ADA during the study period. Treatment-induced ADA = negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result. Treatment-enhanced ADA = a participant with positive ADA result at baseline who has one or more post-baseline titer results that are at least 0.60 t.u. greater than the baseline titer result.
Time Frame: Baseline up to approximately 2 years after last dose (up to approximately 69 months)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 3 | 5 | 10 | 37
Participants
  Baseline prevalence of ADAs: number analyzed (Participants) | 2 | 5 | 10 | 35
  Baseline prevalence of ADAs | 0 | 0 | 0 | 0
  Post baseline incidence of ADAs: number analyzed (Participants) | 3 | 4 | 7 | 37
  Post baseline incidence of ADAs | 0 | 0 | 0 | 0

20. Secondary Outcome: Number of Participants With Anti-therapeutic Antibodies (ATAs) to Polatuzumab Vedotin
Description: The number of participants with positive results for ATAs, also called ADAs against polatuzumab vedotin at baseline and at any of the post-baseline assessment time-points were reported. Number of participants positive for Treatment Emergent ADA = the number of post-baseline evaluable participants determined to have treatment induced ADA or treatment-enhanced ADA during the study period. Treatment-induced ADA = negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result. Treatment-enhanced ADA = a participant with positive ADA result at baseline who has one or more post-baseline titer results that are at least 0.60 t.u. greater than the baseline titer result.
Time Frame: Baseline up to approx. 2 years after the last dose of polatuzumab vedotin (up to approximately 30 months)
Population: Immunogenicity population included all safety-evaluable participants with at least one ADA sample. Due to missing baseline or post-baseline results not every participant was evaluable for baseline prevalence or post-baseline incidence of ADAs. 'Number Analyzed' is the number of participants with data available for analysis at a specified timepoint.
Measure: Count of Participants; unit: Participants
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 15 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
Number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 5 | 10 | 39 | 38
Participants
  Baseline prevalence of ADAs: number analyzed (Participants) | 3 | 4 | 2 | 6 | 3 | 5 | 10 | 38 | 37
  Baseline prevalence of ADAs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 1
  Post baseline incidence of ADAs: number analyzed (Participants) | 3 | 4 | 3 | 6 | 3 | 4 | 7 | 38 | 37
  Post baseline incidence of ADAs | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: From Baseline up to study completion/discontinuation (maximum of 69 months)
Description: The safety-evaluable population was defined as all participants who received at least one dose of any component of the combination.
Arm/Group | Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 15 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL
All-Cause Mortality (participants affected / at risk) | 1/3 | 2/4 | 1/3 | 2/6 | 3/3 | 2/5 | 10/10 | 7/40 | 20/39
Serious Adverse Events (participants affected / at risk) | 3/3 | 2/4 | 2/3 | 3/6 | 0/3 | 0/5 | 4/10 | 26/40 | 19/39
Other Adverse Events (participants affected / at risk) | 3/3 | 4/4 | 3/3 | 6/6 | 3/3 | 5/5 | 9/10 | 40/40 | 37/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL (N=3) | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 1000 mg G in FL (N=4) | Dose-escalation Phase: 1.4 mg Pola + 15 mg L + 1000 mg G in FL (N=3) | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL (N=6) | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL (N=3) | Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL (N=5) | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL (N=10) | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL (N=40) | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL (N=39)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CARDIAC FAILURE (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
PERICARDITIS (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
COLITIS (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRIC HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
LIP SWELLING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PYREXIA (General disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
BRONCHIOLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
COVID-19 PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
EPIDIDYMITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
INJECTION SITE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
LUNG ABSCESS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
NEUTROPENIC SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 2 (2)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
SEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEPTIC SHOCK (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UROSEPSIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANKLE FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FEMUR FRACTURE (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HIP FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
UPPER LIMB FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TUMOUR LYSIS SYNDROME (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
CANCER PAIN (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 1 (1)
BRAIN STEM STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ENCEPHALOPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ISCHAEMIC STROKE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEIZURE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CONFUSIONAL STATE (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
URINARY RETENTION (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOXIA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INTERSTITIAL LUNG DISEASE (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMONITIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PNEUMOTHORAX (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STEVENS-JOHNSON SYNDROME (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dose-escalation Phase: 1.4 mg Pola + 10 mg L + 1000 mg G in FL (N=3) | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 1000 mg G in FL (N=4) | Dose-escalation Phase: 1.4 mg Pola + 15 mg L + 1000 mg G in FL (N=3) | Dose-escalation Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL (N=6) | Dose-escalation Phase: 1.8 mg Pola + 10 mg L + 375 mg R in DLBCL (N=3) | Dose-escalation Phase: 1.8 mg Pola + 15 mg L + 375 mg R in DLBCL (N=5) | Dose-escalation Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL (N=10) | Expansion Phase: 1.4 mg Pola + 20 mg L + 1000 mg G in FL (N=40) | Expansion Phase: 1.8 mg Pola + 20 mg L + 375 mg R in DLBCL (N=39)
ANAEMIA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 1 (2) | 3 (5) | 1 (1) | 2 (3) | 5 (5) | 18 (29) | 14 (22)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (4) | 1 (1)
LYMPHOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (3) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 1 (2) | 2 (9) | 1 (8) | 6 (18) | 2 (7) | 3 (7) | 7 (15) | 26 (117) | 25 (62)
NEUTROPHILIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 1 (1)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 0 (0) | 2 (2) | 1 (3) | 5 (10) | 1 (4) | 1 (6) | 2 (2) | 22 (50) | 10 (18)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
LEFT VENTRICULAR DYSFUNCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TYMPANIC MEMBRANE PERFORATION (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIABETES INSIPIDUS (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPOTHYROIDISM (Endocrine disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DRY EYE (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OCULAR HYPERAEMIA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PERIORBITAL OEDEMA (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
ABDOMINAL PAIN (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 6 (6) | 3 (3)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 4 (5) | 3 (3)
ASCITES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 1 (1) | 7 (10) | 8 (8)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 2 (3) | 2 (2) | 2 (3) | 1 (1) | 1 (1) | 1 (1) | 2 (4) | 17 (24) | 13 (23)
DRY MOUTH (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
DYSPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTRITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HAEMORRHOIDAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
MELAENA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
NAUSEA (Gastrointestinal disorders) | 1 (2) | 1 (2) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 8 (10) | 5 (5)
ODYNOPHAGIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
RECTAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
UMBILICAL HERNIA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 5 (5) | 4 (4)
ASTHENIA (General disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 2 (2) | 7 (12) | 6 (6)
CHILLS (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 2 (2)
FATIGUE (General disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 11 (11) | 6 (6)
FEELING ABNORMAL (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAIT DISTURBANCE (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INFLUENZA LIKE ILLNESS (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4) | 2 (2)
PAIN (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL SWELLING (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 3 (4)
PYREXIA (General disorders) | 2 (3) | 0 (0) | 2 (6) | 3 (3) | 1 (1) | 1 (1) | 1 (2) | 13 (17) | 5 (5)
OCULAR ICTERUS (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CYTOKINE RELEASE SYNDROME (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
HYPOGAMMAGLOBULINAEMIA (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
BRONCHITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CANDIDA INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CLOSTRIDIUM DIFFICILE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
CONJUNCTIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 1 (1)
CYTOMEGALOVIRUS INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GASTROENTERITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2)
INFLUENZA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
LOWER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
NASOPHARYNGITIS (Infections and infestations) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 8 (11) | 2 (2)
ORAL CANDIDIASIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
ORAL HERPES (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (6) | 0 (0)
RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 7 (13) | 3 (3)
RHINITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
SINUSITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (5) | 0 (0)
TONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 1 (2) | 1 (1) | 6 (9) | 2 (2)
UPPER RESPIRATORY TRACT INFECTION BACTERIAL (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
URINARY TRACT INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (5) | 4 (4)
CONTUSION (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FALL (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
INFUSION RELATED REACTION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 17 (19) | 2 (2)
MUSCLE STRAIN (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 1 (2) | 0 (0) | 2 (5) | 1 (1) | 8 (11) | 5 (8)
AMYLASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 1 (4) | 1 (2) | 5 (7) | 4 (8)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 2 (2) | 4 (6) | 0 (0)
BLOOD BILIRUBIN INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (12) | 2 (5)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (10) | 3 (4)
BLOOD GLUCOSE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
BLOOD LACTATE DEHYDROGENASE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 4 (5) | 2 (2)
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (3) | 2 (2)
CARDIAC STRESS TEST ABNORMAL (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CREATININE RENAL CLEARANCE DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CREATININE RENAL CLEARANCE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2) | 2 (2) | 5 (10) | 3 (4)
IMMUNOGLOBULINS DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
LIPASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
TRANSAMINASES INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 8 (8) | 6 (6)
DEHYDRATION (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
GOUT (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 4 (4)
HYPERPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 2 (2) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 4 (7)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (3) | 1 (3) | 0 (0) | 0 (0) | 2 (2) | 2 (6) | 4 (5)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (5) | 1 (1) | 5 (13) | 5 (9)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
HYPOPROTEINAEMIA (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 1 (1) | 2 (3) | 0 (0) | 0 (0) | 0 (0) | 7 (9) | 2 (2)
ARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 5 (5) | 6 (7)
DIASTASIS RECTI ABDOMINIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 5 (7) | 1 (1)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (3)
MYALGIA (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 3 (4) | 0 (0)
NECK PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 2 (2)
SACRAL PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
TENDONITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SQUAMOUS CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
TUMOUR FLARE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
BURNING SENSATION (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
DIZZINESS (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 5 (7) | 3 (4)
DYSGEUSIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 1 (1)
HEAD TITUBATION (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 1 (1) | 0 (0) | 1 (2) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (3)
NEURALGIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 0 (0)
NEUROPATHY PERIPHERAL (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 3 (3) | 3 (3)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
PERIPHERAL MOTOR NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
RESTING TREMOR (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
DEPRESSION (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
INSOMNIA (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
DYSURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 3 (4) | 2 (2)
HAEMATURIA (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
RENAL FAILURE (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
COUGH (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 3 (7) | 0 (0) | 1 (1) | 1 (1) | 10 (11) | 5 (5)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 5 (5) | 1 (1)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (12) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 4 (4) | 1 (1)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 2 (2) | 2 (2)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RHINORRHOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
UPPER-AIRWAY COUGH SYNDROME (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2)
DYSHIDROTIC ECZEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 3 (4) | 0 (0)
PETECHIAE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 4 (4) | 2 (3)
RASH (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 5 (5) | 7 (10)
RASH ERYTHEMATOUS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 3 (4)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
SKIN ULCER (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
URTICARIA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
FLUSHING (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 1 (1)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ORTHOSTATIC HYPOTENSION (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-01-19): https://cdn.clinicaltrials.gov/large-docs/97/NCT02600897/Prot_SAP_000.pdf